CLINICAL TRIAL: NCT06161493
Title: Phase l Study of a BET Inhibitor, ZEN003694, Combined With a PARP Inhibitor, Niraparib in Patients With Metastatic or Recurrent Solid Tumors
Brief Title: ZEN003694 Combined With Niraparib in Patients With Metastatic or Recurrent Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator Discretion
Sponsor: Haider Mahdi (Other)
Collaborators: GlaxoSmithKline (Industry); Zenith Epigenetics (Industry)
Responsible Party: Sponsor-Investigator, Haider Mahdi, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 22-142
Record Dates: First submitted 2023-11-27; First posted 2023-12-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer; Recurrent Solid Tumors
Keywords: BET inhibitor; PARP inhibitor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib (Experimental): ZEN003694: Oral capsules - Starting dose 36 mg Dose escalated to 48 mg, following the mTPI-2/Keyboard design administered orally once daily in 28-day cycles
  Niraparib: Oral tablets - Starting dose 100 mg Dose escalated to 200 mg, following the mTPI-2/Keyboard design administered once daily at the same time as ZEN003694
  Interventions: Drug: ZEN003694; Drug: Niraparib

INTERVENTIONS:
Drug: ZEN003694 — A bromodomain extra-terminal inhibitor (BETi) that blocks a group of proteins called bromodomain and extra-terminal (BET), which may counteract the effect of NSD3 on tumor growth.
Drug: Niraparib — An anti-cancer medication (PARP inhibitor) used for the treatment of epithelial ovarian, fallopian tube, or primary peritoneal cancer .
  Other Names: MK-4827; Zejula

SUMMARY:
This Phase I, open label, dose determining study of oral niraparib in combination with ZEN003694 given daily in 28-day cycles will enroll patients with metastatic or recurrent solid cancer. Dose escalation will follow the mTPI-2/Keyboard design. Eligible patients will receive therapy until disease progression or unacceptable toxicities are experienced.

DETAILED DESCRIPTION:
PARPis impair the repair of single strand DNA breaks leading to double strand DNA breaks especially in patients with defects in the HR pathway. PARP is have been extensively studied in ovarian cancer and are approved for patients with germline or somatic BRCA mutant ovarian cancer after 2-3 lines of chemotherapy. PARPis have been also approved as maintenance therapy in first line and recurrent ovarian cancer after partial or complete response to platinum-based therapy. PARPis have prominent activity in BRCA mutated cancer with lower activity in the BRCA wild type HRD negative ovarian cancer. Approximately 18-24% of ovarian cancer harbor somatic or germline BRCA mutation and 50% harbor alteration in the homologous recombination (HR) pathway.

Further, PARPi therapy is frequently associated with PARPi resistance. Therefore, there is a need to reverse PARPi resistance and enhance response to PARPi in PARPi resistant ovarian cancer. Recently, significant pre-clinical evidence has shown that BETi's synergize with PARPi's through downregulation of the transcription of several HR genes. It is hypothesized that BETi may suppress HR and enhance non-homologous end joining thereby sensitizing HR-proficient cancer cells to PARP inhibition, and also BETi has been described to reverse PARPi resistance. To test this hypothesis, this Phase I trial will test the combination of niraparib and ZEN003694 in recurrent or metastatic solid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) status 0 or 1
* Pathologically documented recurrent or metastatic solid tumor who progressed on standard of care therapy or for whom standard of care does not exist.
* Prior PARPi therapy is allowed
* Have had no more than 5 prior cancer therapy treatment regimens, of which a maximum of 4 were cytotoxic chemotherapy or DNA-damaging agents like PARPi-containing regimens
* Measurable disease per RECIST 1.1
* Known BRCA1/2 status or willing to be tested
* Adequate laboratory parameters at Screening
* Treated females patients not breastfeeding, pregnant or of childbearing potential, or permanently sterile or who are post-menopausal (no menses for at least 1 year without an alternative medical cause and FSH levels in the post-menopausal range)
* Ability to swallow capsules and comply with study procedures
* Ability to sign informed consent form prior to initiation of any study procedures.
* Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study enrollment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable with evidence of no disease progression for 6 months.

Exclusion Criteria:

* Current or anticipated use of medications known to be strong inhibitors or inducers of CYP3A4 or substrates of CYP1A2 with narrow therapeutic windows. Strong inhibitors, inducers or substrates must be discontinued at least 7 days prior to the first administration of study drug.
* Current or anticipated use within 7 days prior to the first administration of study drug, or during the study, of strong P-gp inhibitors.
* Use of oral Factor Xa inhibitors (i.e., rivaroxaban, apixaban, betrixaban, edoxaban otamixaban, letaxaban, eribaxaban) and Factor IIa inhibitors (i.e., dabigatran). Low molecular weight heparin is allowed
* Radiation to >25% of the bone marrow
* Treatment with a bone-targeted radionuclide within 6 weeks of first dose of study drug
* Have previously received an investigational BET inhibitor (including previous participation in studies with Zenith drug, ZEN003694)
* QTcF interval > 470 msec
* Insufficient recovery from prior treatment-related toxicities except for alopecia, fatigue and Grade 2 neuropathy
* Non-healing wound, ulcer or bone fracture (not including a pathological bone fracture caused by a pre-existing pathological bone lesion)
* Brain metastases not adequately treated and/or clinically stable (at the discretion of the Investigator) for at least 6 months prior to the start of study treatment.
* Known impaired cardiac function or clinically significant cardiac disease such as uncontrolled supraventricular arrhythmia, ventricular arrhythmia requiring therapy, or congestive heart failure (New York Heart Association functional class III or IV)
* Myocardial infarction or unstable angina within 6 months prior to the first administration of study drug
* Known myelodysplastic syndrome
* Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active central nervous system disease, active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, or any other condition that could compromise safety or the patient's participation in the study
* Impairment of gastrointestinal function that may significantly alter the absorption of ZEN003694 or niraparib
* Other known active cancer requiring therapy at time of study entry or that progressed or required treatment within 3 years prior to starting study drug (except for skin basal cell carcinoma or squamous cell carcinoma or in situ cervical cancer)
* Prior history with PRES
* Hypersensitivity to the active substance of to any of the excipients, including tartrazine in the capsule formulation.
* Patients with not adequately controlled hypertension despite adequate medical treatment.
* History of infection with (screening tests not required): human immunodeficiency virus; hepatitis B virus with currently active disease defined as hepatitis B surface antigen (HBsAg) positivity; or hepatitis C virus unless previously treated and viral load is undetectable except following situations:

  * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of enrollment are eligible for this trial.
  * Patients with a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection are allowed to be included if: participant on a stable dose of antiviral therapy, HBV viral load below the limit of quantification. HCV viral load below the limit of quantification.
* Major surgery other than diagnostic surgery, dental surgery or stenting within 4 weeks prior to the first administration of study drug
* Concurrent participation in another clinical investigational treatment trial
* Any other reason that in the opinion of the Investigator would prevent the patient from completing participation or following the study schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-related Adverse Events (AE) and Serious Adverse Events (SAE) | Up to 36 months (study population)
  Frequency and severity of adverse events (AE) per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0. The maximum grade for each toxicity type will be recorded for each patient.
Maximum Tolerated Dose (MTD) / Recommended Phase 2 Dose (RP2D) | Up to 12 months (study population)
  Frequency of dose-limiting toxicities (DLTs) (AEs leading to discontinuation of treatment).
  The mTPI-2/Keyboard design is a Bayesian interval dose determining design. The target toxicity rate for the MTD for this combination therapy is defined at 0.30 with an acceptable toxicity probability interval (0.25, 0.35). The MTD is selected based on the dose estimate closest to the target toxicity rate, and the recommend phase II dose will be determined based on the MTD and all available safety and PK data.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Up to 30 days
  Maximum observed concentration (Cmax) in blood taken from patients treated with ZEN003694 combined with niraparib.
Pharmacodynamics (PD) | Up to 30 days
  Area under the serum concentration-time curve (AUC) in blood taken from patients treated with ZEN003694 combined with niraparib.
Objective response rate (ORR) by RECIST 1.1 | Up to 6 years (study population)
  Proportion of participants achieving a best response of CR or PR per RECIST v1.1, at each dose level. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Duration of Response | Up to 6 years (study population)
  Time from start of treatment to disease progression or death in patients who achieve Complete Response (CR) or Partial Response (PR) (whichever is recorded first) per RECIST v1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free survival (PFS) | Up to 6 years (study population)
  Median number of months from start of treatment to the date of disease progression or death from any cause. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall survival (OS) | Up to 6 years (study population)
  Median length of time from start of treatment that patients remain alive.

CONTACTS AND LOCATIONS:
Overall Officials: Haider S Mahdi, MD, Principal Investigator — UPMC Magee Women's Hospital, UPMC Hillman Cancer Center
Locations (1):
- UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No